CLINICAL TRIAL: NCT03314142
Title: Short-term Effects of Bran Size on Glycemic Responses in Normal Weight Healthy Adults
Brief Title: Effects of Bran Size on Glycemic Responses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agricultural University of Athens (Other)
Responsible Party: Principal Investigator, Aimilia Papakonstantinou, Lecturer in Nutrition and Metabolism, Agricultural University of Athens
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 1256
Record Dates: First submitted 2017-10-02; First posted 2017-10-19 (Actual); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Potential Abnormality of Glucose Tolerance; Appetitive Behavior
Keywords: blood glucose; bran particle size; glucemic index
MeSH Terms: conditions — Appetitive Behavior | interventions — Glucose

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Glucose as reference food (Experimental): Ten healthy, normal weight subjects (male: 7, female: 3) after 10-14 hr fast, consumed 50g available carbohydrate from white bread and glucose, two times, in different weeks as reference foods along with 250ml water; and 50g available carbohydrates from bread enriched with coarse wheat bran (CB), bread enriched with fine wheat bran (obtained by milling the coarse bran) (FB) and the FB in which 10% of the flour was substituted with carob seed flour (CSFB), tested once, in different weeks along with 250ml water. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120min. The first glucose sample was taken exactly 15min after the first bite of food or drink.
  Interventions: Other: Glucose as reference food; Other: White bread as reference food; Other: Bread enriched with coarse wheat bran; Other: Bread enriched with fine wheat bran; Other: Bread enriched with fine wheat bran and carob seed flour
- White bread as reference food (Experimental): Ten healthy, normal weight subjects (male: 7, female: 3) after 10-14 hr fast, consumed 50g available carbohydrate from white bread and glucose, two times, in different weeks as reference foods along with 250ml water; and 50g available carbohydrates from bread enriched with coarse wheat bran (CB), bread enriched with fine wheat bran (obtained by milling the coarse bran) (FB) and the FB in which 10% of the flour was substituted with carob seed flour (CSFB), tested once, in different weeks along with 250ml water. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120min. The first glucose sample was taken exactly 15min after the first bite of food or drink.
  Interventions: Other: Glucose as reference food; Other: White bread as reference food; Other: Bread enriched with coarse wheat bran; Other: Bread enriched with fine wheat bran; Other: Bread enriched with fine wheat bran and carob seed flour
- Bread enriched with coarse wheat bran (Experimental): Ten healthy, normal weight subjects (male: 7, female: 3) after 10-14 hr fast, consumed 50g available carbohydrate from white bread and glucose, two times, in different weeks as reference foods along with 250ml water; and 50g available carbohydrates from bread enriched with coarse wheat bran (CB), bread enriched with fine wheat bran (obtained by milling the coarse bran) (FB) and the FB in which 10% of the flour was substituted with carob seed flour (CSFB), tested once, in different weeks along with 250ml water. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120min. The first glucose sample was taken exactly 15min after the first bite of food or drink.
  Interventions: Other: Glucose as reference food; Other: White bread as reference food; Other: Bread enriched with coarse wheat bran; Other: Bread enriched with fine wheat bran; Other: Bread enriched with fine wheat bran and carob seed flour
- Bread enriched with fine wheat bran (Experimental): Ten healthy, normal weight subjects (male: 7, female: 3) after 10-14 hr fast, consumed 50g available carbohydrate from white bread and glucose, two times, in different weeks as reference foods along with 250ml water; and 50g available carbohydrates from bread enriched with coarse wheat bran (CB), bread enriched with fine wheat bran (obtained by milling the coarse bran) (FB) and the FB in which 10% of the flour was substituted with carob seed flour (CSFB), tested once, in different weeks along with 250ml water. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120min. The first glucose sample was taken exactly 15min after the first bite of food or drink.
  Interventions: Other: Glucose as reference food; Other: White bread as reference food; Other: Bread enriched with coarse wheat bran; Other: Bread enriched with fine wheat bran; Other: Bread enriched with fine wheat bran and carob seed flour
- Bread enriched with fine wheat and carob (Experimental): Ten healthy, normal weight subjects (male: 7, female: 3) after 10-14 hr fast, consumed 50g available carbohydrate from white bread and glucose, two times, in different weeks as reference foods along with 250ml water; and 50g available carbohydrates from bread enriched with coarse wheat bran (CB), bread enriched with fine wheat bran (obtained by milling the coarse bran) (FB) and the FB in which 10% of the flour was substituted with carob seed flour (CSFB), tested once, in different weeks along with 250ml water. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120min. The first glucose sample was taken exactly 15min after the first bite of food or drink.
  Interventions: Other: Glucose as reference food; Other: White bread as reference food; Other: Bread enriched with coarse wheat bran; Other: Bread enriched with fine wheat bran; Other: Bread enriched with fine wheat bran and carob seed flour

INTERVENTIONS:
Other: Glucose as reference food — Ten subjects (male: 7, female: 3) consumed 50g glucose diluted in 250ml water, tested three times, in different weeks, within 5-10min. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120min.
Other: White bread as reference food — Ten subjects (male: 7, female: 3) consumed 50g available carbohydrates from white bread along with 250ml water, tested twice, in different weeks, within 5-10min. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120min.
Other: Bread enriched with coarse wheat bran — Ten subjects (male: 7, female: 3) consumed 50g available carbohydrates from bread enriched with coarse wheat bran along with 250ml water, tested once, in different weeks, within 5-10min. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120 min.
Other: Bread enriched with fine wheat bran — Ten subjects (male: 7, female: 3) consumed 50g available carbohydrates from bread enriched with fine wheat bran (obtained by milling of the coarse bran) along with 250ml water, tested once, in different weeks, within 5-10min. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120 min.
Other: Bread enriched with fine wheat bran and carob seed flour — Ten subjects (male: 7, female: 3) consumed 50g available carbohydrates from bread enriched with fine wheat bran (obtained by milling of the coarse bran) in which 10% of the flour was substituted with carob seed flour (CSFB) along with 250ml water, tested once, in different weeks, within 5-10min. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120 min.

SUMMARY:
This study investigated the effects of bran's particle size on glycemic responses

DETAILED DESCRIPTION:
This study aimed at 1. to determine the GI and GL of three breads and 2. to investigate the effects of bran's particle size on postprandial glycemic response in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-smoking, non-diabetic men and women, individuals with normal body mass index (BMI; between 18.5 and 24.9 kg/m2)

Exclusion Criteria:

* severe chronic disease (e.g. coronary heart disease, diabetes mellitus, kidney or liver conditions, endocrine conditions)
* gastrointestinal disorders
* pregnancy
* lactation
* competitive sports
* alcohol or drug dependency

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Capillary blood glucose responses | 2 hours
  Clinically useful change in blood glucose, defined as the restoration of glucose within normal limits during the 2hr glucose tolerance test.

SECONDARY OUTCOMES:
Subjective appetite ratings | 2 hours
  Useful change in subjective appetite using visual analogue scales (VAS, 100 mm, given in the form of booklet, one scale per page) before and 2hr after consumption of four different bread types.

CONTACTS AND LOCATIONS:
Overall Officials: Emilia Papakonstantinou, PhD, Principal Investigator — Agricultural University of Athens
Locations (1):
- Agricultural University of Athens, Athens, Greece

IPD SHARING:
Plan to Share IPD: No